CLINICAL TRIAL: NCT04092101
Title: Low Nicotine Content Cigarettes in Vulnerable Populations: Opioid Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); National Institute on Drug Abuse (NIDA) (NIH); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Stacey C. Sigmon, Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CHRMS19-0130; U54DA036114-06 (NIH)
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Tobacco Use Disorder
Keywords: Biomarkers of Exposure; Compensatory Smoking; Nicotine Dependence; Reduced Nicotine Cigarettes; Affective Disorders; Tobacco Withdrawal; Vulnerable Populations; E-Cigarettes
MeSH Terms: conditions — Tobacco Use Disorder; Mood Disorders; Vaping | interventions — Tobacco Products; Electronic Nicotine Delivery Systems

STUDY DESIGN:
Intervention Model Description: Randomized parallel groups research design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind dosing of tobacco cigarette nicotine levels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RC 1 only (Experimental): Research Cigarettes #1
  Interventions: Other: Cigarettes with varying nicotine content
- RC 2 only (Experimental): Research Cigarettes #2
  Interventions: Other: Cigarettes with varying nicotine content
- RC 2 + EC 1 (Experimental): Research Cigarettes #2 plus E-cigarettes #1
  Interventions: Other: Cigarettes with varying nicotine content; Other: E-Cigarettes
- RC 2 + EC 2 (Experimental): Research Cigarettes #2 plus E-cigarettes #2
  Interventions: Other: Cigarettes with varying nicotine content; Other: E-Cigarettes

INTERVENTIONS:
Other: Cigarettes with varying nicotine content — 1) Altering the nicotine content of the tobacco research cigarette
Other: E-Cigarettes — 1) Altering the availability of e-cigarettes; 2) Altering option to personalize the e-liquid in the e-cig condition
  Arms: RC 2 + EC 1; RC 2 + EC 2

SUMMARY:
Prevalence of smoking among individuals with opioid use disorder (OUD) is six-fold that of the general US adult population. The mortality rate of opioid-dependent smokers is four times that of opioid-dependent nonsmokers, and their response to smoking cessation interventions is notoriously poor. A national policy of reducing the nicotine content of cigarettes has the potential to be an effective method of reducing tobacco use prevalence, dependence, and related adverse health outcomes. Controlled trials in the general smoker population have demonstrated that switching smokers to low nicotine content cigarettes results in reductions in cigarettes per day (CPD), dependence and tobacco toxicant exposure, with few adverse consequences. The investigators believe that the impact of reduced nicotine standards on use of combusted cigarettes in this population will be moderated considerably by other tobacco market conditions including (1) availability of alternative sources of non-combusted nicotine, and (2) whether these alternatives are available under conditions that optimize their appeal. The investigators hypothesize the same for other vulnerable populations as well, but achieving significant reductions in use of combusted cigarettes in smokers with OUD seems especially unlikely in the absence of readily available and appealing alternative sources of non-combusted nicotine.

The goal of the proposed trial is to experimentally model whether increased availability and appeal of an alternative, non-combusted source of nicotine (e-cigarettes) will enhance the effectiveness of a reduced nicotine standard for cigarettes in smokers with OUD. Additionally, the investigators will test whether allowing participants to personalize the favor of the e-liquid alters any moderating effects their availability may have on tobacco cigarette smoking.

Daily smokers who are receiving methadone or buprenorphine treatment will be recruited at University of Vermont and Johns Hopkins University.

The investigators will study two research cigarettes referred to here as RC1 and RC2. One of these cigarettes will be a normal nicotine content cigarette and the other will be a reduced nicotine content cigarette. Investigators will study two e-cigarette conditions referred to here as EC1 and EC2. Both e-cigarette conditions will involve the same commercially available devices and same nicotine-containing e-liquid, but in one condition that e-liquid will be available only in tobacco flavor while in the other condition that e-liquid will be available in multiple flavors from which participants can choose based on personal taste preference. Participants will be assigned to one of the following four study conditions: (1) RC1 only; (2) RC2 only; (3) RC2 + EC1; (4) RC2 + EC2.

Participants will be asked to use only their assigned study products for 16 weeks. Outcome measures include total CPD, cigarette demand assessed by behavioral economics-based purchase tasks, craving, withdrawal, psychiatric symptoms, breath carbon monoxide (CO), and biomarkers of tobacco toxicant exposure.

ELIGIBILITY:
Inclusion Criteria:

* Maintained on opioid medication
* 21 to 70 years old

Exclusion Criteria:

* Not maintained on opioid medication
* Under 21 years old
* Over 70 years old

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2020-10-18 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacey C. Sigmon, Ph.D., Principal Investigator — University of Vermont
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Shirley Plucinski, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Higgins ST, Sigmon SC, Tidey JW, Heil SH, Gaalema DE, Lee DC, DeSarno MJ, Klemperer EM, Menson KE, Cioe PA, Plucinski S, Wiley RC, Orr E. Reduced Nicotine Cigarettes and E-Cigarettes in High-Risk Populations: 3 Randomized Clinical Trials. JAMA Netw Open. 2024 Sep 3;7(9):e2431731. doi: 10.1001/jamanetworkopen.2024.31731. PMID 39240566

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RC 1 Only | RC 2 Only | RC 2 + EC 1 | RC 2 + EC 2
Started | 83 | 85 | 74 | 84
Completed | 67 | 66 | 57 | 70
Not Completed | 16 | 19 | 17 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RC 1 Only | RC 2 Only | RC 2 + EC 1 | RC 2 + EC 2 | Total
Number analyzed (Participants) | 83 | 85 | 74 | 84 | 326
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.77 (10.98) | 39.85 (9.28) | 41.51 (12.39) | 39.38 (10.59) | 40.09 (10.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 69 | 50 | 59 | 243
  Male | 18 | 16 | 24 | 25 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 3 | 2 | 12
  Not Hispanic or Latino | 79 | 82 | 71 | 82 | 314
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 6 | 9 | 9 | 34
  White | 67 | 70 | 61 | 68 | 266
  More than one race | 4 | 7 | 1 | 4 | 16
  Unknown or Not Reported | 1 | 1 | 3 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 83 | 85 | 74 | 84 | 326
Population [Count of Participants; unit: Participants] — Vulnerable population subgroups
  Females with lower educational level : Daily female smokers of reproductive age (21-44 years) with lower educational level (< Associate's degree)
  Opioid Use Disorder: Daily smokers on methadone or buprenorphine treatment for Opioid Used Disorder
  Affective Disorders: Daily smokers with past year MDD, dysthymic disorder, generalized anxiety disorder, post-traumatic stress disorder, obsessive-compulsive disorder, or panic disorder
  Participants
    Females with lower educational level | 20 | 23 | 16 | 21 | 80
    Opioid Use Disorder | 19 | 19 | 17 | 19 | 74
    Affective disorders | 44 | 43 | 41 | 44 | 172
Educational level [Count of Participants; unit: Participants]
  <High school | 9 | 4 | 3 | 14 | 30
  High school graduate, equivalency, or some college | 51 | 57 | 46 | 47 | 201
  Associate's degree | 8 | 11 | 13 | 11 | 43
  ≥College graduate | 15 | 13 | 12 | 12 | 52
Marital status [Count of Participants; unit: Participants]
  Married | 8 | 15 | 17 | 11 | 51
  Never married | 49 | 47 | 36 | 48 | 180
  Divorced, separated, or widowed | 26 | 23 | 21 | 25 | 95
Primarily smokes mentholated cigarettes [Count of Participants; unit: Participants] | 32 | 35 | 31 | 33 | 131
Cigarettes smoked per day [Mean (Standard Deviation); unit: cigarettes per day] | 16.42 (8.02) | 18.44 (9.47) | 17.86 (9.11) | 16.90 (8.85) | 17.40 (8.87)
Urine cotinine level [Mean (Standard Deviation); unit: ng/mL] | 4499.25 (3120.20) | 5235.67 (3251.28) | 5156.57 (4150.44) | 5293.33 (3799.45) | 5043.55 (3680.12)
Breath CO level [Mean (Standard Deviation); unit: ppm] | 20.90 (14.02) | 19.30 (12.39) | 21.03 (13.38) | 20.66 (13.44) | 20.46 (13.28)
Age started smoking regularly [Mean (Standard Deviation); unit: years] | 16.61 (3.97) | 15.92 (3.91) | 16.24 (3.84) | 16.79 (5.15) | 16.39 (4.26)
FTND total score [Mean (Standard Deviation); unit: scores on a scale] — Fagerstrom Test for Nicotine Dependence
  In scoring the Fagerstrom Test for Nicotine Dependence, the three yes/no items are scored 0 (no) and 1 (yes). The three multiple-choice items are scored from 0 to 3.
  The items are summed to yield a total score of 0-10.
  Classification of dependence based on total score:
  0-2 Very low 3-4 Low 5 Moderate 6-7 High 8-10 Very high
  scores on a scale | 5.12 (2.24) | 5.31 (2.20) | 5.26 (2.31) | 4.70 (2.07) | 5.09 (2.21)
Used other tobacco products, past 30 days [Count of Participants; unit: Participants] | 5 | 4 | 5 | 9 | 23
Used e-cigarettes, past 30 days [Count of Participants; unit: Participants] | 13 | 11 | 5 | 13 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Cigarettes Smoked Per Day
Description: Cigarettes per day will be assessed for use of cigarettes with different nicotine content.
Time Frame: 16 weeks
Population: Participants who completed week 16 of study
Measure: Least Squares Mean (Standard Error); unit: cigarettes per day
Arm/Group | RC 1 Only | RC 2 Only | RC 2 + EC 1 | RC 2 + EC 2
Number analyzed (Participants) | 67 | 66 | 57 | 70
cigarettes per day | 22.54 (1.59) | 14.32 (1.32) | 11.76 (1.18) | 7.63 (0.90)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | RC 1 Only | RC 2 Only | RC 2 + EC 1 | RC 2 + EC 2
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/85 | 1/74 | 0/84
Serious Adverse Events (participants affected / at risk) | 9/83 | 4/85 | 4/74 | 2/84
Other Adverse Events (participants affected / at risk) | 71/83 | 74/85 | 62/74 | 72/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RC 1 Only (N=83) | RC 2 Only (N=85) | RC 2 + EC 1 (N=74) | RC 2 + EC 2 (N=84)
Psychiatric disorders - Other (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Esophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pregnancy, puerperium, and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death NOS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury, poisoning, and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RC 1 Only (N=83) | RC 2 Only (N=85) | RC 2 + EC 1 (N=74) | RC 2 + EC 2 (N=84)
OASIS Score Increase (Psychiatric disorders) | 32 (51) | 31 (43) | 31 (42) | 31 (40)
BDI Category Increase (Psychiatric disorders) | 29 (51) | 29 (40) | 26 (34) | 25 (41)
Psychiatric disorders (Psychiatric disorders) | 27 (53) | 28 (43) | 19 (27) | 24 (37)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 23 (38) | 27 (44) | 18 (40) | 18 (35)
General disorders and administration (General disorders) | 18 (25) | 24 (27) | 16 (20) | 22 (27)
Infections and infestations (Infections and infestations) | 16 (17) | 23 (24) | 8 (11) | 10 (13)
Nervous system disorders (Nervous system disorders) | 7 (8) | 18 (23) | 15 (19) | 10 (11)
Gastrointestinal disorders (Gastrointestinal disorders) | 9 (14) | 17 (25) | 14 (20) | 17 (23)
Vascular disorders (Vascular disorders) | 10 (13) | 13 (15) | 8 (10) | 16 (30)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 11 (14) | 16 (16) | 7 (7) | 12 (12)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 6 (7) | 4 (7) | 4 (4) | 5 (8)
Surgical and medical procedures (Surgical and medical procedures) | 2 (2) | 3 (3) | 5 (5) | 4 (4)
Cardiac disorders (Cardiac disorders) | 4 (6) | 2 (4) | 3 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT04092101/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT04092101/ICF_001.pdf